CLINICAL TRIAL: NCT06162195
Title: The ACTIVE Trial: A Prospective Randomised Control Trial Of The H1 Implant Versus Total Hip Replacement
Acronym: ACTIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Embody Orthopaedic Limited (Industry)
Collaborators: Imperial College London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 327954
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Hip; Inflammatory Arthritis
Keywords: Hip; Resurfacing; Ceramic
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Intervention Model Description: Randomisation will be performed using variable block randomisation with block sizes of 4, 6 and 8, with a 1:1 allocation to the 2 groups, with stratification across sites. This will ensure approximately equal numbers across groups and approximately the same number per group at each site (to control for differences in the trial population because of environmental, social and demographic factors), while allowing different total numbers at each site. It will also ensure that at any given time, the numbers in each group will be approximately equal, allowing the interim analyses to take place. The randomisation will be managed by the contract research organisation (CRO) via an electronic data capture (EDC) system, which uses a validated randomisation algorithm. Once a patient has been consented, they will be assigned to a treatment group according to the pre-determined order inside the block. Stratification by site is recommended for multi-centre studies.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients, clinical assessors and data analysts will be blinded to the intervention each patient has received for the 24 month post-operative period. The surgeon, operating theatre team, radiographic analysts and CRO cannot be blinded but will not be involved in the care of the patient after the intervention unless the patient requires revision surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The H1 Implant (Experimental): Cementless, ceramic-on-ceramic hip resurfacing arthroplasty (HRA) device.
  Interventions: Device: The H1 Implant
- Cementless total hip replacement (Active Comparator): Cementless ceramic-on-poly or ceramic-on-ceramic total hip replacement
  Interventions: Device: Cementless total hip replacement

INTERVENTIONS:
Device: The H1 Implant — Patients allocated to The H1 Implant arm will be implanted with the H1 Implant which is a cementless, ceramic hip resurfacing device.
  Arms: The H1 Implant
Device: Cementless total hip replacement — Patients allocated to cementless total hip replacement arm will be implanted with a cementless ceramic-on-poly or ceramic-on-ceramic total hip replacement
  Arms: Cementless total hip replacement

SUMMARY:
The goal of this randomised controlled trial is to compare the success of two types of hip replacement in patients with hip arthritis. The main question it aims to answer is whether a new type of hip replacement (called a hip resurfacing) can be as successful as an existing hip replacement (called a total hip replacement). Patients will be given either the new hip resurfacing or the existing total hip replacement and researchers will compare their function, complication rate and physical activity.

DETAILED DESCRIPTION:
The H1 Implant is a cementless, ceramic hip resurfacing arthroplasty (HRA) device. The intended purpose of the H1 Implant is to provide an artificial substitute for a disease-damaged hip joint to replace the articulating surfaces of the hip while preserving the underlying femoral head and natural femoral neck. This is standard for a resurfacing hip prosthesis. This study will randomise patients to receive either The H1 Implant or a primary cementless ceramic-on-poly or ceramic-on-ceramic total hip replacement (THR). Composite clinical success (CCS) scores, physical activity levels and patient reported outcome measures (PROMs) will be compared for the two groups. The primary objective of the study is to determine whether the H1 Implant is non-inferior to cementless THR in terms of CCS. The key secondary objective is to determine whether the H1 Implant is superior compared to cementless THR in terms of physical activity and PROMs. Other secondary objectives are to compare the H1 Implant and THR with respect to: safety, through collection of all device-related, operative site-related and systemic adverse events; and noise generation, through patient survey.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires unilateral primary hip arthroplasty due to primary osteoarthritis, osteoarthritis secondary to e.g. trauma, avascular necrosis or developmental hip dysplasia, or inflammatory arthritis.
* Patient is willing to comply with study requirements.
* Patient plans to be available through 10 years postoperative follow-up.

Exclusion Criteria:

* Patient has a BMI greater than 40 kg/m².
* Patient has active infection or sepsis (treated or untreated).
* Patient has insufficient bone stock at the hip (>1/3 necrosis of the femoral head or large and multiple cysts) or in general as in severe osteopenia or osteoporosis (t-score < -2.5 as measured with BMD).
* Patient is not skeletally mature.
* Patient meets the contraindication criteria of the control device.
* Patient already has another lower limb arthroplasty or arthrodesis or will require a further lower limb arthroplasty or arthrodesis within the subsequent 2 years.
* Patient lacks capacity to consent.
* Patient is unable to understand the native language of the country where their procedure is taking place

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Composite clinical success (CCS) | 24 months post-operatively
  The primary outcome is "composite clinical success". This is a binary outcome measure. Patients are deemed to have achieved CCS if they meet all of the following criteria at the 24 month timepoint:
  * Modified Harris Hip Score ≥80.
  * No revision or pending revision.
  * Acetabular radiolucencies: not in all zones.
  * Femoral radiolucencies: not in all zones.
  * Absence of subsidence/migration of the acetabular or femoral component >5mm with clinical findings.
  * Absence of specific adverse device effects (ADEs) that are pre-cursors to revision of the device, namely:
    * Bone breakage around the implanted component(s) (periprosthetic fracture).
    * Breakage of the device component.
    * Device movement/migration of clinical consequence as defined by associated clinical findings as: a limp; leg length discrepancy; and restricted range of motion.
    * Dislocation of the hip joint.

SECONDARY OUTCOMES:
Physical Activity | 6 months, 12 months and 24 months post-operatively
  Average daily minutes of activity and mean bouted daily moderate-vigorous physical activity (MVPA), minutes
Physical Activity | Pre-operatively, 6 months, 12 months and 24 months post-operatively
  Physical performance assessment: number of chair stands in 30 seconds and time taken to perform stair climb test
Physical Activity | Pre-operatively, 6 months, 12 months and 24 months post-operatively
  Hip Outcome Score (HOS) Questionnaire
Physical Activity | Pre-operatively, 6 months, 12 months and 24 months post-operatively
  UCLA (University of California Los Angeles) Activity Score
Noise | 6 weeks, 6 months, 12 months and 24 months post-operatively
  Noise questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Justin Cobb, Prof, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No